CLINICAL TRIAL: NCT05785221
Title: Exploratory Personalized Lifestyle Intervention on Metabolic Homeostasis in Overweight or Obese Chinese Population
Brief Title: Energy Metabolism Profiles Over Weight-loss and Eating Responses
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xu Lin, Principal Investigator, Chinese Academy of Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HIAS-LIMH-202302
Record Dates: First submitted 2023-03-01; First posted 2023-03-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Homeostasis; Metabolism and Nutrition Disorder; Healthy; Obesity
Keywords: Metabolic homeostasis; Healthy; Lifestyle intervention
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Comparators (Placebo Comparator): They will receive general lifestyle and nutritional education.
  Interventions: Behavioral: General lifestyle and nutritional education
- Overweight/Obese Group (Experimental): They will receive personalized nutritional and lifestyle weight reduction intervention including dietary advice, behavior guidance and nutritional and lifestyle education by dietitian and physicians.
  Interventions: Behavioral: Personalized nutritional and lifestyle weight reduction intervention

INTERVENTIONS:
Behavioral: General lifestyle and nutritional education — Participants will receive general dietary advice, behavior guidance and nutritional and lifestyle education based on dietary guidelines.
  Arms: Healthy Comparators
Behavioral: Personalized nutritional and lifestyle weight reduction intervention — Participants will receive personalized dietary advice, behavior guidance and nutritional and lifestyle education by dietitian and physicians. APP-connected wearable devices will be utilized to monitor their dietary intakes, physical activities and sleep conditions and APP-connected scale will be used to monitor their weight changes during interventions.
  Arms: Overweight/Obese Group

SUMMARY:
This is an exploratory controlled before-after study, which involves 112 participants, of whom 28 are with normal weight and 84 are overweight or obese. Twelve weeks of caloric-restriction dietary intervention will be conducted in the overweight or obese participants. Before and after the 12-week intervention, metabolic health will be characterized by metabolic homeostasis, determined via comprehensive measurements of dynamic postprandial metabolic responses to a standardized mixed macronutrient tolerance test (75 g glucose, 60 g fat, 20 g protein) in a whole-room indirect calorimeter. The objectives of this study are

1. to characterize dynamic metabolic response elicited by acute nutritional and acute exercise challenges,
2. to elucidate biological mechanisms underlying inter-individual heterogeneity in these responses,
3. to predict prospective weight loss over the intervention using heterogeneous metabolic responses to acute challenges

DETAILED DESCRIPTION:
The objectives of this study are 1) to characterize dynamic metabolic response elicited by acute nutritional and acute exercise challenges, 2) to elucidate biological mechanisms underlying inter-individual heterogeneity in these responses, and 3) to predict prospective weight loss over the intervention using heterogeneous metabolic responses to acute challenges.

In this study, 84 overweight or obese participants (BMI ≥ 24 kg/m2) and 28 normal weight participants (18.5 ≤ BMI<24 kg/m2) will be recruited and receive 12-week caloric-restriction dietary or weight maintenance interventions. Before and after the 12-week interventions, metabolic homeostasis will be used to characterize metabolic health and to be determined using comprehensive measurements of dynamic changes in postprandial metabolic responses (including energy metabolism, multiple clinical biomarkers, metabolomic signatures, gut microbiota, genetic signatures etc.) after standardized mixed macronutrient tolerance test (75 g glucose, 60 g fat and 20 g protein) in whole room indirect calorimeter under both resting and exercise conditions. In addition, data from dietary intake, anthropometric measurements, body composition, psychosocial measures, behavior questionnaires and 14-day continuous glucose monitoring will also be collected to characterize metabolic homeostasis. During the interventions, participants will receive personalized dietary advice, behavior guidance and nutritional and lifestyle education by dietitian and physicians. APP-connected wearable devices will be utilized to monitor their dietary intakes, physical activities and sleep conditions, and an application-connected scale will be used to monitor their weight changes during interventions. The study's protocol has been approved by the Ethics Committee of Sir Run Run Shaw Hospital.

ELIGIBILITY:
Inclusion Criteria:

* 20-70 years of age, inclusive
* BMI ≥ 24kg/m2
* Not in other clinical studies currently or in the past three months

Exclusion Criteria:

* Fasting glucose >7.0mmol/L or diagnosed diabetes or taking insulin or other blood glucose-lowering drugs
* Blood pressure > 160/100 mmHg; diagnosed phase II or III hypertension or cannot decrease SBP under 160mmHg after anti-hypertension drugs
* Fasting blood TG≥ 5.7 mmol/L or fasting LDL-C≥ 4.9 mmol/L or cannot control TG < 5.7 mmol/L or LDL-C < 4.9 mmol/L after taking lipid lowering drugs
* Pregnant or lactating
* Attempting to change body weight in the past 3 months
* Use of antibiotic in the preceding 3 months for 3-serial days
* Use of estrogen therapy or hormonal drugs in the preceding 6 months
* Smokers
* History of alcohol abuse or other substance abuse (Alcohol abuse is defined as regular alcohol consumption > 40 g/day for females or > 80 g/day for males)
* Severe renal disease or liver disease
* Severe gastrointestinal diseases
* Surgical events preceding 1 year (except appendicitis or hernia surgery)
* Severe cardiovascular or cerebrovascular diseases
* Implantation of heart stent or any device containing metal material
* Cancer or receiving radiotherapy and chemotherapy within 5 years
* Hyperthyroidism or hypothyroidism
* Suffering from AIDS, hepatitis A, hepatitis B and other infectious diseases
* Claustrophobia
* Physical disability
* Any mental disorders or current use of antidepressants
* Cognitive disability

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Fasting and postprandial energy metabolic response at baseline and post-intervention | Baseline and Week 12
  Energy metabolism is characterized by four primary indicators: energy expenditure (EE), respiratory quotient (RQ), carbohydrate oxidation rate (CarbOx), and fat oxidation rate (FatOx).
  EE denotes the rate of energy expenditure per minute (typically expressed in kcal/min).
  RQ, defined as the ratio of carbon dioxide produced to oxygen consumed (VCO₂/VO₂), reflects whole-body substrate utilization.
  CarbOx and FatOx represent the respective oxidation rates of carbohydrate and fat, quantifying the contribution of each macronutrient to total energy production.

SECONDARY OUTCOMES:
Change from Baseline in Body Weight at 12 Weeks | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention. Weight will be assessed by Seca-255 (ScalesGalore).
Change from Baseline in Body Mass Index at 12 Weeks | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention. Weight and height will be assessed by Seca-255 (ScalesGalore).
Change from Baseline in Waist Circumference at 12 Weeks | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention. Waist circumference will be assessed by Seca-201(ScalesGalore).
Change from Baseline in Hip Circumference at 12 Weeks | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention. Waist circumference will be assessed by Seca-201(ScalesGalore).
Change from Baseline in Blood Pressure at 12 Weeks | Baseline and Week 12
  The change of systolic and diastolic blood pressures between the baseline and after 12-week lifestyle intervention. Both systolic pressure and diastolic pressure will be assessed using electronic blood pressure monitor (Omron J750).
Change from Baseline in Heart Rate at 12 Weeks | Baseline and Week 12
  The change of systolic and diastolic blood pressures between the baseline and after 12-week lifestyle intervention. Heart rate will be assessed using Omron J750.
Change from Baseline in Body Composition at 12 Weeks | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention. Body composition will assessed using dual energy x-ray absorptiometry (DXA) (GE).
Change from Baseline in Energy Expenditure at 12 Weeks | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention. Energy expenditure will be assessed using whole room indirect calorimeter.
Change from Baseline in Respiratory Quotient at 12 Weeks | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention. Respiratory quotient will be assessed using whole room indirect calorimeter.
Change from Baseline in Glucose Homeostasis at 12 Weeks | Baseline and Week 12
  The change between the baseline and after 12-week lifestyle intervention. Glucose homeostasis will be assessed by Continuous Glucose Monitoring (FreeStyle Libre).
Change from Baseline in Glucose at 12 Weeks | Baseline and Week 12
  The dynamic change of glucose from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in C-peptide at 12 Weeks | Baseline and Week 12
  The dynamic change of C-peptide from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in Insulin Indices at 12 Weeks | Baseline and Week 12
  The dynamic change of insulin indices from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in Lipid Parameters at 12 Weeks | Baseline and Week 12
  The dynamic change of lipid parameters from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in Protein and Amino Acids Metabolites at 12 Weeks | Baseline and Week 12
  The dynamic change from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in Inflammatory Biomarkers and Cytokines at 12 Weeks | Baseline and Week 12
  The dynamic change from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in Gastrointestinal Hormones at 12 Weeks | Baseline and Week 12
  The dynamic change in gastrointestinal hormones from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in Cell Adhesion Molecules at 12 Weeks | Baseline and Week 12
  The dynamic change in cell adhesion molecules from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in Adipokines at 12 Weeks | Baseline and Week 12
  The dynamic change in adipokines from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention.
Change from Baseline in Metabolomics at 12 Weeks | Baseline and Week 12
  The dynamic change in metabolomics including profiling of free fatty acids and other metabolites from 0 to 30, 60, 120, 180, 240, 300 minutes pre- and post-oral mixed-nutrient dietary challenge between the baseline and after 12-week lifestyle intervention. Metabolomics will be measured by LC-MS.
Single nucleotide polymorphism (SNPs) | Baseline
  Mutations at specific sites will be detected by gene chip.
Gut microbiota 16S rDNA sequencing | Baseline and Week 12
  Gut microbiota 16S rDNA will be sequenced and community composition will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, PhD, Principal Investigator — Institute for Nutritional Sciecnes, CAS; Hangzhou Institute for Advanced Study, UCAS
Locations (1):
- Hangzhou Institute for Advanced Study, University of Chinese Academy of Sciences, Hangzhou, Zhejiang, China